CLINICAL TRIAL: NCT00474994
Title: A Multicenter Phase II Study of Continuous Dosing of Sunitinib (Sutent®, SU11248) in Non-GIST Sarcomas
Brief Title: Sunitinib in Treating Patients With Metastatic, Locally Advanced, or Locally Recurrent Sarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-054; P30CA008748 (NIH); MSKCC-07054; PFIZER-MSKCC-07054
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-12

CONDITIONS: Adult Malignant Fibrous Histiocytoma of Bone; Desmoid Tumor; Endometrial Cancer; Ovarian Cancer; Sarcoma; Small Intestine Cancer
Keywords: chondrosarcoma; recurrent osteosarcoma; localized adult malignant fibrous histiocytoma of bone; metastatic adult malignant fibrous histiocytoma of bone; recurrent adult malignant fibrous histiocytoma of bone; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Kaposi sarcoma; recurrent uterine sarcoma; adult leiomyosarcoma; adult malignant fibrous histiocytoma; adult rhabdomyosarcoma; dermatofibrosarcoma protuberans; stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma; ovarian sarcoma; uterine leiomyosarcoma; stage III uterine sarcoma; stage IV uterine sarcoma; desmoid tumor; adult angiosarcoma; recurrent adult soft tissue sarcoma; uterine carcinosarcoma; endometrial stromal sarcoma; fibrosarcomatous osteosarcoma; chondrosarcomatous osteosarcoma; adult alveolar soft-part sarcoma; adult epithelioid sarcoma; adult extraskeletal chondrosarcoma; adult extraskeletal osteosarcoma; adult fibrosarcoma; adult malignant hemangiopericytoma; adult malignant mesenchymoma; adult neurofibrosarcoma; adult synovial sarcoma; adult desmoplastic small round cell tumor; adult liposarcoma; anaplastic osteosarcoma; mixed osteosarcoma; small intestine leiomyosarcoma; osteoblastic osteosarcoma; telangiectatic osteosarcoma; classic Kaposi sarcoma; immunosuppressive treatment related Kaposi sarcoma; AIDS-related Kaposi sarcoma
MeSH Terms: conditions — Histiocytoma, Malignant Fibrous; Desmoid Tumors; Endometrial Neoplasms; Ovarian Neoplasms; Sarcoma; Chondrosarcoma; Osteosarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Sarcoma, Kaposi; Leiomyosarcoma; Rhabdomyosarcoma; Dermatofibrosarcoma; Hemangiosarcoma; Sarcoma, Endometrial Stromal; Sarcoma, Alveolar Soft Part; Chondrosarcoma, Extraskeletal Myxoid; Fibrosarcoma; Hemangiopericytoma, Malignant; Malignant mesenchymal tumor; Neurofibrosarcoma; Sarcoma, Synovial; Desmoplastic Small Round Cell Tumor; Liposarcoma; Bone Neoplasms; AIDS-related Kaposi sarcoma | interventions — Sunitinib

ARMS (3):
- Group A (Experimental): Vascular connective tissue neoplasms, leiomyosarcoma, dermatofibrosarcoma protuberans (DFSP), desmoid tumors. Sunitinib 37.5 mg daily continuously; one cycle is 28 days. Restaging: after every 2 cycles until after 6 cycles, when restaging will be decreased to once every 3 cycles.
  Interventions: Drug: sunitinib malate
- Group B (Experimental): High grade undifferentiated pleomorphic sarcoma (includes the older designation malignant fibrous histiocytoma [MFH]) and other non-GIST connective tissue tumors; may include carcinosarcomas.Sunitinib 37.5 mg daily continuously; one cycle is 28 days. Restaging: after every 2 cycles until after 6 cycles, when restaging will be decreased to once every 3 cycles.
  Interventions: Drug: sunitinib malate
- Group C (Experimental): Chordomas. Sunitinib 37.5 mg daily continuously; one cycle is 28 days. Restaging: after every 2 cycles until after 6 cycles, when restaging will be decreased to once every 3 cycles.
  Interventions: Drug: sunitinib malate

INTERVENTIONS:
Drug: sunitinib malate

SUMMARY:
RATIONALE: Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well sunitinib works in treating patients with metastatic, locally advanced, or locally recurrent sarcomas.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate (complete response and partial response) in patients with metastatic, locally advanced, or locally recurrent non-gastrointestinal stromal tumor sarcomas treated with sunitinib malate.

Secondary

* Determine the 16- and 24-week progression-free survival rate (complete response, partial response, and stable disease) in patients treated with this drug.
* Determine the overall survival in patients treated with this drug.
* Correlate clinical response with changes in soluble angiogenesis mediator levels in patients treated with this drug.
* Determine the tumor maximum standardized uptake values by fludeoxyglucose F 18-PET scan in patients treated with this drug.

OUTLINE: This is a multicenter study. Patients are stratified by neoplastic subtype (vascular connective tissue neoplasms, leiomyosarcoma, dermatofibrosarcoma protuberans, chordoma, or desmoid tumors vs high-grade undifferentiated pleomorphic sarcoma [i.e., malignant fibrous histiocytoma (including myxofibrosarcoma)], or other nongastrointestinal connective tissue tumors [including carcinosarcomas]).

Patients receive oral sunitinib malate once daily on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed connective tissue neoplasm, including any of the following neoplastic subtypes:

  * Vascular connective tissue neoplasms
  * Leiomyosarcoma
  * Dermatofibrosarcoma protuberans
  * Chordoma
  * Desmoid tumors
  * High-grade undifferentiated pleomorphic sarcoma (e.g., malignant fibrous histiocytoma [including myxofibrosarcoma])
  * Carcinosarcomas (e.g., malignant mixed Müllerian tumors)
  * Giant hemangiomata
  * Kaposi sarcoma
* Metastatic, locally advanced, or locally recurrent disease
* Measurable disease

  * Tumor lesions in a previously irradiated area may be considered measurable provided there is evidence of growth that cannot be attributed to necrosis or bleeding
* No gastrointestinal stromal tumor sarcomas
* Prior standard neoadjuvant or adjuvant systemic therapy required for patients with the following diagnoses:

  * Rhabdomyosarcoma
  * Osteosarcoma
  * Ewing sarcoma
* No untreated brain metastases, spinal cord compression, or evidence of symptomatic brain metastases or leptomeningeal disease as documented on screening CT scan or MRI

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 mg/dL
* PT and INR ≤ 1.5
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine ≤ 1.5 mg/dL
* Calcium ≤ 12 mg/dL
* Blood glucose < 150 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception prior to, during, and for 28 days after completion of study therapy
* Other malignancies allowed provided sarcoma is the primary disease requiring systemic therapy
* Able to swallow oral medications
* No other disease or illness within the past 6 months, including any of the following:

  * Myocardial infarction
  * Severe or unstable angina
  * Coronary or peripheral artery bypass graft
  * Symptomatic congestive heart failure
  * Cerebrovascular accident or transient ischemic attack
  * Pulmonary embolism
* No evidence of a bleeding diathesis
* No ongoing cardiac dysrhythmias > grade 2
* No uncontrolled hypertension, defined as blood pressure > 150/100 mm Hg despite optimal medical therapy
* Left ventricular ejection fraction ≥ 50% by echocardiogram or MUGA scan
* No psychiatric illness or social situation that would preclude study compliance
* No pre-existing thyroid abnormality, defined as abnormal thyroid function tests despite medication
* No prolonged QTc interval (i.e., QTc > 450 msec for males or QTc > 470 msec for females) on baseline EKG
* No hemorrhage ≥ grade 3 in the past 4 weeks

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* No prior sunitinib malate
* No more than 3 prior cytotoxic chemotherapy regimens for metastatic disease

  * Adjuvant chemotherapy for sarcoma completed > 1 year prior to study entry is not considered a line of prior treatment
* At least 2 weeks since prior cytotoxic chemotherapy
* At least 6 weeks since prior carmustine or mitomycin C
* At least 1 week since prior biological therapy or small molecule kinase inhibitors
* At least 3 weeks since prior radiotherapy (except for palliative radiotherapy to specific sites)

  * Prior palliative radiotherapy allowed provided it is considered medically necessary and there are other target lesions to assess
* More than 4 weeks since prior major surgery
* Concurrent major surgery allowed provided study drug is stopped 2 weeks before surgery and resumed 2 weeks after surgery
* Concurrent palliative radiotherapy (e.g., focal radiotherapy to a bony metastasis for relieving bone pain) allowed
* No other concurrent investigational drugs
* No concurrent participation in another clinical trial
* No concurrent therapeutic anticoagulation (e.g., warfarin)

  * Prophylactic anticoagulation (i.e., low-dose warfarin) of venous or arterial access devices allowed provided requirements for PT and INR are met
* No other concurrent approved or investigational anticancer agents or treatment, including chemotherapy, biological response modifier therapy, hormonal therapy, or immunotherapy

  * Concurrent hormone replacement therapy for adrenal insufficiency allowed
* No concurrent antiepileptic drugs (e.g., phenytoin, carbamazepine, or phenobarbital)
* No concurrent rifampin, theophylline, ketoconazole, or Hypericum perforatum (St. John's wort)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary L. Keohan, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Robert Maki, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- [Result] George S, Merriam P, Maki RG, Van den Abbeele AD, Yap JT, Akhurst T, Harmon DC, Bhuchar G, O'Mara MM, D'Adamo DR, Morgan J, Schwartz GK, Wagner AJ, Butrynski JE, Demetri GD, Keohan ML. Multicenter phase II trial of sunitinib in the treatment of nongastrointestinal stromal tumor sarcomas. J Clin Oncol. 2009 Jul 1;27(19):3154-60. doi: 10.1200/JCO.2008.20.9890. Epub 2009 May 18. PMID 19451429

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib (Sutent®, SU11248) in Non-GIST Sarcomas: Sunitinib (Sutent®, SU11248) in Non-GIST Sarcomas
Period: Overall Study
Arm/Group | Sunitinib (Sutent®, SU11248) in Non-GIST Sarcomas
Started | 53
Completed | 48
Not Completed | 5
Not completed — Patient Not treated | 1
Not completed — Patient evaluable for toxicity only | 3
Not completed — Patient found to be ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib (Sutent®, SU11248) in Non-GIST Sarcomas
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 45
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response
Description: as assessed by RECIST criteria
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Sunitinib (Sutent®, SU11248) in Non-GIST Sarcomas
Number analyzed (Participants) | 48
participants
  Partial Response (PR) | 1
  Stable Disease (SD) | 21
  Progression of Disease (POD) | 26

ADVERSE EVENTS:
Arm/Group | Sunitinib (Sutent®, SU11248) in Non-GIST Sarcomas
Serious Adverse Events (participants affected / at risk) | 9/53
Other Adverse Events (participants affected / at risk) | 37/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib (Sutent®, SU11248) in Non-GIST Sarcomas (N=53)
Death not associated with CTCAE term- Death NOS (General disorders) | 1 (1)
Death not associated with CTCAE term-Disease progression NOS (General disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (2)
Pain - Abdomen NOS (General disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Pneumothorax (Gastrointestinal disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (2)
Thrombosis/thrombus/embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ulcer, Duodenum (Gastrointestinal disorders) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib (Sutent®, SU11248) in Non-GIST Sarcomas (N=53)
AST, SGOT (Blood and lymphatic system disorders) | 3 (3)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 6 (6)
Gastrointestinal, other (Gastrointestinal disorders) | 3 (3)
Hemoglobin (Blood and lymphatic system disorders) | 5 (5)
Hypertension (Cardiac disorders) | 9 (9)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 14 (14)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3)
Mucositis (Clincal exam)- Oral cavity (General disorders) | 7 (7)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 15 (15)
Platelets (Blood and lymphatic system disorders) | 7 (7)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes